CLINICAL TRIAL: NCT05249998
Title: Improving Care of Prader-Willi Syndrome : Evaluation of a New Care Program Combining Adapted Physical Activity, Nutrition and Therapeutic Education
Acronym: APHYNET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: APHP200143
Record Dates: First submitted 2021-10-15; First posted 2022-02-22 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Prader-Willi Syndrome; Obesity
Keywords: Prader Willi Syndrome; Therapeutic Education; Adapted Physical Activity; Nutrition
MeSH Terms: conditions — Prader-Willi Syndrome; Obesity | interventions — Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional group (Experimental): Patients will receive the usual care, with the intervention of the multidisciplinary team which defines with the patient the objectives of the stay and the inter-stay period, without "specific therapeutic education" on adapted physical activity, nutrition and eating behaviour.
  Interventions: Other: Program combing APA, Nutrition, and Therapeutic Education
- Standard care group (No Intervention): Patients will benefit from the activities already proposed as part of the usual practice and in addition a multidisciplinary staff will take place in order to interpret the assessments of the patients included and to direct the patients according to their phenotypic profile towards the different programmes of adapted physical activity.

INTERVENTIONS:
Other: Program combing APA, Nutrition, and Therapeutic Education — Patients will benefit from the activities already proposed as part of the usual practice and in addition a multidisciplinary staff will take place in order to interpret the assessments of the patients included and to direct the patients according to their phenotypic profile towards the different programmes of adapted physical activity.
  Arms: Interventional group

SUMMARY:
Prader-Willi syndrome (PWS) is a rare and complex genetic disease characterized by hypothalamic-pituitary axis dysfunction combining eating disorders associated with hyperphagia and satiety deficiency, mild intellectual deficit and behavioral disorders. This disease requires continuous management through specific therapeutic education to prevent metabolic and cardiorespiratory complications related to obesity. Physical activity must therefore be regular, adapted to the disability, taking into account cognitive deficits and behavioral disorders.

The Unit of Care and Rehabilitation, of the Hôpital Marin d'Hendaye, receives patients with PWS or other obesity from rare causes, at a rate of 1 to 2 annual stays of 1 to 2 months, which allow the regulation of somatic disorders and the initiation of weight loss. However, the difficulty is to keep a stable weight curve between stays. Only 20% of patients over the last 2 years managed to stabilize or decrease their BMI during the 6 months following their hospitalization.

The proposed study aims to evaluate an innovative and individualized care program combining Physical activity, Nutrition and therapeutic education for adults with PWS who will be admitted to the hospital for 5 weeks.

We hypothesize that this program will allow to stabilize or decrease the BMI of patients at 6 months after hospitalization by inducing a behavioral change in terms of physical activity and eating behavior.

We will conduct a randomized controlled trial on 128 patients who will participate in this program, or will benefit from standard care.

DETAILED DESCRIPTION:
Main objective :

Evaluate the effectiveness at 6 months of an intensified and individualised care programme combining theoretical and practical therapeutic education workshops on adapted physical activity, nutrition and eating behaviour (i.e. intervention) during hospitalisation, compared to usual care (i.e. control).

The assessment will be done by comparing the proportion of patients stabilizing or decreasing their BMI at 6 months after the end of the stay (M7) in the 2 groups (intervention/control).

Secondary objectives:

During hospitalization:

To evaluate, compared to the usual care, the impact of the intervention on :

1. The evolution of physical capacities,
2. The evolution of metabolic criteria and metabolic and cardio-respiratory risk factors,
3. The evolution of eating behaviour,
4. Adherence to the program during hospitalization.

At 3 and 6 months after hospitalization :

Evaluate the impact of the intervention on :

1. The evolution of weekly physical activity at home,
2. The evolution of eating behaviour at home,
3. Reaching the personalized objective set for the inter-stay.

At 6 months after hospitalization:

Evaluate, in comparison with the usual management, the impact of the intervention on the evolution of metabolic criteria and metabolic and cardio-respiratory risk factors during a consultation at the hospital in their reference center.

ELIGIBILITY:
Inclusion Criteria:

* Patient between 18 and 60 years old Patient with genetically confirmed PWS
* Admitted for a 5-week stay in the Hendaye rehabilitation care unit
* Patient or legal guardian (tutor or curator) who has given written informed consent to participate in the study
* With the presence of an external relay available to coordinate the patient's journey during the protocol: family or educational referent (home)
* Affiliated with French social security except patient under AME (State medical aid)

Exclusion Criteria:

* Decompensation of a cardiorespiratory or psychiatric pathology in the 3 months prior to inclusion that required hospitalisation
* Patients whose condition may interfere with their optimal participation in the study (e.g., severe behavioural problems preventing participation in group workshops)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2021-11-06 (Actual); Primary Completion 2024-05-04 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Change in Body Mass Index (BMI) | week 4
Change in Body Mass Index (BMI) | week 7

SECONDARY OUTCOMES:
six minute walking test (6MWT) | week 4
Forced Vital Capacity | baseline and week 4
Maximum Volume Expired in the 1st Second | baseline and week 4
Prospective assessment of clinical features before and after Adapted Physical Activity Program | baseline and week 4
  Weight in kilograms, Height in meters to calculate Body Mass Index (BMI) in kg/m^2
Difference of CRP dosage between before and after Adapted Physical Activity Program | baseline and week 4
  CRP measured before and after Adapted Physical Activity Program : difference between these two dosages
Difference of Glycated hemoglobin (Hba1C) between before and after Adapted Physical Activity Program | baseline and week 4
  Glycated hemoglobin (Hba1C) measured before and after Adapted Physical Activity Program : difference between these two dosages
Difference of fasting blood glucose between before and after Adapted Physical Activity Program | baseline and week 4
  fasting blood glucose level measured before and after Adapted Physical Activity Program : difference between these two dosages
Difference of cholesterol between before and after Adapted Physical Activity Program | baseline and week 4
  Cholesterol measured before and after Adapted Physical Activity Program : difference between these two dosages
Difference of Glycemy between before and after Adapted Physical Activity Program | baseline and week 4
  Glycemy measured before and after Adapted Physical Activity Program : difference between these two dosages
Difference of transaminases between before and after Adapted Physical Activity Program | baseline and week 4
  Transaminases measured before and after Adapted Physical Activity Program : difference between these two dosages
Difference of Gamma GT between before and after Adapted Physical Activity Program | baseline and week 4
  Gamma GT measured before and after Adapted Physical Activity Program : difference between these two dosages
Difference of Alkaline phosphatase between before and after Adapted Physical Activity Program | baseline and week 4
  Alkaline phosphatase measured before and after Adapted Physical Activity Program : difference between these two dosages
Difference of urea between before and after Adapted Physical Activity Program | baseline and week 4
  Urea measured before and after Adapted Physical Activity Program : difference between these two dosages
Difference of creatinine between before and after Adapted Physical Activity Program | baseline and week 4
  creatinine measured before and after Adapted Physical Activity Program : difference between these two dosages
Difference of albumin between before and after Adapted Physical Activity Program | baseline and week 4
  albumin measured before and after Adapted Physical Activity Program : difference between these two dosages
RELIME : REal LIfe Meal Evaluation score | baseline and week 4
  This score is devided in 3 under-scores which are:
  * "eating behavior score" scale of 0 to 30
  * "general behavior score" scale of 0 to 20
  * "social behavior score" scale of 0 to 16 The final score is on a scale of 0 to 66. 0 is the minimum and the best score. 66 is the maximum and worst score.
Adhesion Grid Scores | baseline and week 4
  This score is devided in 2 scores which are :
  "adhesion" on a scale of 0 to 2 "motivation" on a scale of 0 to 2
  The final score is the addition of them on a scale of 0 to 4. The minimum and worst score is 0. The maximum and best score is 4.
Ricci & Gagnon self-questionnaire | baseline, Month 4, Month 7
  This score is on a scale of 0 to 45, 0 is the minimum and worst score and 45 the maximum and worst score of physical activity.
  Score under 18 means "inactive" Score between 18 and 35 means "active" Score superior to 35 means "very active"
Hyperphagia Questionnaire | baseline, Month 4, Month 7
  This score is devided in 3 under-scores which are :
  * "hyperphagic behavior" score on a scale of 5 to 25
  * "hyperphagic drive" score on a scale of 4 to 20
  * "hyperphagic severity" score on a scale of 2 to 10 The final score is on a scale of 11 to 55. 11 is the minimum and best score. 55 is the maximum and worst score.
Goal Attainment Scaling | baseline, Month 4, Month 7
  Goal Attainment Scaling (GAS) is a method for writting personalized evaluation scales in order to quantify progress towards defined goals.
  The GAS methodology consists of:
  * defining an rehabilitation goal with the patient
  * choosing an observable behavior that reflects the degree of goal attainment
  * assessing the patient's initial level (pre- intervention) with respect to the goal
  * defining five goal attainment levels , ranging from "no change" (-2) to "a much better than expected outcome" (+2)
  * Evaluating the patient after the set time frame and determine the GAS score between -2 and +2
  A five point scale is used :
  " -2 " is the baseline ; " -1 " represents progression to the goal without goal attainment ; " 0 " is the expected level after intervention ; " +1 " is represent a better outcome than expected ; " +2 " is the best possible outcometha t could have been expected to the goal
  Scores between " 0 " and " +2 " indicate that the patient has achieved the objective
Weight | Month 2, Month 3, Month 4, Month 5, Month 6, Month 7

CONTACTS AND LOCATIONS:
Overall Officials: Hélène PASTRE, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service diététique Hôpital Marin d'Hendaye- AP-HP, Hendaye, France

IPD SHARING:
Plan to Share IPD: No